CLINICAL TRIAL: NCT05521503
Title: Cardiac Biopsy Collection Repository and Database
Brief Title: Biopsy Collection and Repository Database
Acronym: BICARD
Status: Recruiting | Type: Observational
Sponsor: Kenneth S. Campbell (Other)
Responsible Party: Sponsor-Investigator, Kenneth S. Campbell, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 73647
Record Dates: First submitted 2022-08-20; First posted 2022-08-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During this study, tissue samples (blood, urine and/or myocardial tissue) will be used to help identify trends in biomarkers and other information for patients with Cardiac Amyloidosis and other Cardiovascular conditions. No clinically important information that could be used by the subject will be identified. Therefore, the results of these studies will not be shared with the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biological specimens: Biological specimens taken from cardiovascular procedures

SUMMARY:
Use samples procured from patients to improve understanding of molecular, cellular, and tissue-level processes produced by a variety of cardiac diseases and therapeutic interventions.

DETAILED DESCRIPTION:
This is a prospective study enrolling patients referred for or undergoing cardiovascular procedures or treatment at the University of Kentucky. The study aims to facilitate the discovery of novel diagnostic biomarkers and therapeutic targets and improve the pathophysiological understanding of cardiac conditions.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing evaluation of a cardiac condition or receiving a right heart catheterization with biopsy clinically indicated who are at least 18 years of age.

Exclusion Criteria:

* Patients without a cardiovascular or amyloidosis diagnosis, under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing evaluation of a cardiac condition or receiving a right heart catheterization with biopsy clinically indicated who are at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Discover and quantify the concentration of novel diagnostic and prognostic biomarkers | 12/21/2021-12/31/2030
  Use biospecimens procured from patients with cardiac conditions to identify diagnostic surrogate biomarkers using discovery proteomics. In Cardiac Amyloidosis, the serum levels will be compared between confirmed ATTR and non-ATTR heart failure patients and a diagnostic threshold will be established. The research aims to advance understanding of cardiac diseases and to support the development of improved therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Campbell, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States